CLINICAL TRIAL: NCT06435910
Title: Engineered Dendritic Cell Vaccines for Remission Maintenance in Multiple Myeloma Patients
Brief Title: Engineered Dendritic Cell Vaccines for Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: The No.2 Clinical Hospital of the Ministry of Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-24002
Record Dates: First submitted 2024-05-14; First posted 2024-05-30 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma or Plasmacytoma
Keywords: MM; CAR T; DC vaccine
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCvac cells to treat MM (Experimental)
  Interventions: Biological: DC vaccines

INTERVENTIONS:
Biological: DC vaccines — Antigen-presenting and immune modifying DCvacs to treat MM

SUMMARY:
The purpose of this study is to determine the feasibility, safety, and efficacy of dendritic cell (DC) vaccines in the treatment of multiple myeloma (MM) or plasmacytoma based on immune-modified DC vaccines (DCvac). This approach is aimed to achieve prolonged maintenance of remission in multiple myeloma or plasmacytoma patients.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a plasma cell malignancy, characterized by the aberrant occupation of bone marrow with malignant plasma cells, and the destruction of bones together with the production of abnormal immunoglobulins. The clinical symptoms and signs can be manifested through various mechanisms. At present, the therapeutic drugs for MM include glucocorticoid, cytotoxic drugs, immunosuppressants, protease inhibitors, monoclonal antibodies and cell therapies including hematopoietic stem cell transplantation (HSCT). Among them, immunotherapy has been proven to be a revolutionary treatment with great potential of producing long term cure.

In the past decades, adoptively transferred T cells modified with chimeric antigen receptors (CARs) have demonstrated high effectiveness, and the CAR-T therapy has changed the treatment paradigm for many hematological malignancies. Currently, several antibody-based therapies and a few BCMA-based CAR-T cell therapies have been approved for MM treatment. However, in many MM patients, the disease may still relapse after extensive immunotherapies including auto- and allo-HSCT. We have previously reported a DC-based immune activation strategy against MM in a preclinical study. This study proposes to apply the individual patients' MM tumor antigen-based DCs as vaccines (DCvac) to booster anti-myeloma immunity, in order to prevent disease relapse. The MM patients who have achieved very good partial or complete remission will be treated with multiple DCvacs to achieve a prolonged remission without disease recurrence.

This trial protocol will inject DCvacs to MM or plasmacytoma patients who have been treated with a combination of anti-cancer regimens, including CAR-T cell therapy, and who have achieved partial or complete disease remission. The DCvacs are patient's own DCs which are immune modified to present target antigens and to activate anti-cancer immunity. The aim of this study is to evaluate the feasibility, safety, and efficacy of the innovative MM patient-based DC vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with multiple myeloma or plasmacytoma
* Very good partial or complete remission (CR) after prior combination therapies.
* Expected survival > 12 weeks
* Adequate venous access for blood withdrawal or apheresis, and no other contraindications for blood withdrawal
* Voluntary informed consent is given with willingness to continue follow up

Exclusion Criteria:

* Pregnant or lactating women
* Uncontrolled active infection
* HIV or active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids; the use of inhaled steroids is not exclusionary

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2027-07-11 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of DC injection | 1 Month
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Clinical response | 1 year
  Anti-tumor activity of the DCvacs by examination of anti-cancer immunity by measurement of tumor burden

CONTACTS AND LOCATIONS:
Locations (2):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China
- The Regional Hematology Center in Clinical Hospital No. 2 of the Ministry of Health, Vladivostok, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han S, Wang B, Cotter MJ, Yang LJ, Zucali J, Moreb JS, Chang LJ. Overcoming immune tolerance against multiple myeloma with lentiviral calnexin-engineered dendritic cells. Mol Ther. 2008 Feb;16(2):269-79. doi: 10.1038/sj.mt.6300369. Epub 2007 Dec 11. PMID 18071334
- [Background] Ayed AO, Chang LJ, Moreb JS. Immunotherapy for multiple myeloma: Current status and future directions. Crit Rev Oncol Hematol. 2015 Dec;96(3):399-412. doi: 10.1016/j.critrevonc.2015.06.006. Epub 2015 Jun 28. PMID 26153389